CLINICAL TRIAL: NCT03337789
Title: Efficacy of Polygonatum Sibiricum on Sleep Quality Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Jieun Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSE
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Healthy Adults With Subjective Sleep Complaints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polygonatum sibiricum (Experimental)
  Interventions: Dietary Supplement: Polygonatum sibiricum
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Polygonatum sibiricum — Polygonatum sibiricum 800mg, 30-60 minutes before sleep, once a day for 4 weeks
  Arms: Polygonatum sibiricum
Dietary Supplement: Placebo — Placebo 800mg, 30-60 minutes before sleep, once a day for 4 weeks
  Arms: Placebo

SUMMARY:
This study aims to investigate the efficacy and safety of Polygonatum sibiricum for sleep quality improvement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers who are between the ages of 20 and 65
* Experienced any of the following sleep problems, at least more than once a week for more than 2 months: 1) difficulty in falling asleep or staying asleep; 2) waking up at dusk and not being able to fall asleep again; 3) not feeling refreshed even after getting some sleep.

Exclusion Criteria:

* Diagnosed with insomnia assessed with a structured interview and sleep scale measurements
* Possibility of drug-induced sleep disorders due to current intake of medication (i.e., corticosteroid, statin, etc)
* Had taken sleeping pills (i.e., zolpidem, benzodiazepine) during the past 2 months
* Diagnosed with any major medical or neurological disorders assessed during medical history taking, physical examination or experimental tests.
* Diagnosed with any axis 1 psychiatric disorders (depressive disorder, bipolar disorder, alcohol dependence, schizophrenia) evaluated with a structured instrument
* A history of traumatic brain injury with loss of consciousness, or any contraindications to MRI (i.e., claustrophobia, metallic foreign devices in body)
* Had taken psychotropic drugs within the past 3 months before study participation
* Allergic to polygonatum sibiricum or experienced side effects after consumption of any product containing polygonatum sibiricum
* Participated in another clinical trial or took other medications during the period that may influence the results of this clinical trial
* Currently taking contraceptive pills
* Planning for pregnancy during the period of study participation, currently pregnant or breastfeeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline subjective sleep quality at 4 weeks assessed by Pittsburgh Sleep Quality Index | Baseline and week 4
Chagne from baseline physical activity at 4 weeks assessed by actigraph | Baseline and week 4
Change from baseline objective sleep quality at 4 weeks assessed by polysomnography | Baseline and week 4

SECONDARY OUTCOMES:
Change from baseline cognitive functions at 4 weeks assessed by the neuropsychological test battery | Baseline and week 4
Change from baseline depressive symptom levels at 4 weeks assessed by the Hamilton Depression Rating Scale | Baseline and week 4
  Scale name: Hamilton Depression Rating Scale
  / Range of total score: 0 - 52 (Higher scores represent more severe depressive symptoms.)
Change from baseline anxiety symptom levels at 4 weeks assessed by the Hamilton Anxiety Rating Scale | Baseline and week 4
  Scale name: Hamilton Anxiety Rating Scale
  / Range of total score: 0 - 56 (Higher scores represent more severe anxiety symptoms.)
Change from baseline brain structure, function, and metabolism at 4 weeks assessed by computational analysis of magnetic resonance imaging data | Baseline and week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University, Seoul, South Korea